CLINICAL TRIAL: NCT04963738
Title: An Open-label, Single-dose, Parallel-group Study to Evaluate the Effect of Renal Impairment on the Pharmacokinetics of JNJ-73763989 in Adult Participants
Brief Title: A Study of JNJ-73763989 in Adult Participants With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR109019; 2021-001048-85 (EudraCT Number); 73763989HPB1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-07-08; First posted 2021-07-15 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1: JNJ-73763989 (Experimental): Participants with moderate renal impairment will receive a single subcutaneous (SC) injection of JNJ-73763989 on Day 1.
  Interventions: Drug: JNJ-73763989
- Group 2: JNJ-73763989 (Experimental): Participants with severe renal impairment or end-stage renal disease (ESRD) will receive a single SC injection of JNJ-73763989 on Day 1.
  Interventions: Drug: JNJ-73763989
- Group 3: JNJ-73763989 (Experimental): Participants with normal renal function will receive a single SC injection of JNJ-73763989 on Day 1.
  Interventions: Drug: JNJ-73763989

INTERVENTIONS:
Drug: JNJ-73763989 — JNJ-73763989 will be administered as a single SC injection.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of a single subcutaneous (SC) dose of JNJ-73763989 in adult participants with renal impairment compared with healthy participants with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Must have stable renal function defined as a less than (<) 20 percent (%) change in serum creatinine concentrations between screening and Day -1
* Concomitant medications should be stable for the previous 1 month and throughout the duration of the study
* Women, except for postmenopausal women, must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and urine (beta-hCG) pregnancy test on Day -1
* Must sign an informed consent form (ICF) indicating they understand the purpose of, and procedures required for the study and are willing to participate in the study
* Participants with kidney disease without dialysis using benzodiazepines, tricyclic antidepressants, and prescription opiates with a positive urine test for drugs prescribed by their physician may be included following prior discussion with the sponsor

Exclusion Criteria:

* Have kidney disease requiring dialysis
* Renal transplants, systemic lupus erythematosus, or participant with malignancy
* Known allergies, hypersensitivity, or intolerance to JNJ-73763989 or its excipients
* Received an experimental drug (including investigational vaccines) or used an experimental medical device within 1 month or within a period less than 10 times the drug's half-life, whichever is longer, before the administration of the study drug is scheduled
* Preplanned surgery or procedures that would interfere with the conduct of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of JNJ-73763989 | Predose, up to 72 hours postdose (up to Day 4)
  Plasma samples will be analyzed to determine concentrations of JNJ-73763989 (as the 2 triggers JNJ-73763976 and JNJ-73763924) using a validated and qualified method.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 42 days
  AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with AEs by Severity Grades | Up to 42 days
  Number of participants with AEs by severity grade will be reported. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Number of Participants with Abnormalities in Clinical Laboratory Tests, Electrocardiograms (ECGs), Vital Signs and Physical Examination | Up to 42 days
  Number of participants with abnormalities in clinical laboratory tests (including hematology, blood biochemistry, blood coagulation, urinalysis, and urine chemistry), ECGs, vital signs (such as blood pressure, pulse/heart rate, body temperature [tympanic]) and physical examination (including height, body weight, and skin examination) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency